CLINICAL TRIAL: NCT00481091
Title: A Phase 1/2a Study Evaluating the Safety, Pharmacokinetics, and Efficacy of ABT-263 in Subjects With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: A Study of ABT-263 in Participants With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M06-873; 2007-002143-25 (EudraCT Number)
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Results first posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia (CLL); Navitoclax; ABT-263; Cancer
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — navitoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Navitoclax 14/21 Day Cycle: 10 mg (Experimental): Navitoclax 10 mg administered for 14 consecutive days followed by 7 days off drug to complete a 21-day cycle.
  Interventions: Drug: ABT-263
- Navitoclax 14/21 Day Cycle: 110 mg (Experimental): Navitoclax 110 mg administered for 14 consecutive days followed by 7 days off drug to complete a 21-day cycle.
  Interventions: Drug: ABT-263
- Navitoclax 14/21 Day Cycle: 200 mg (Experimental): Navitoclax 200 mg administered for 14 consecutive days followed by 7 days off drug to complete a 21-day cycle.
  Interventions: Drug: ABT-263
- Navitoclax 14/21 Day Cycle: 250 mg (Experimental): Navitoclax 250 mg administered for 14 consecutive days followed by 7 days off drug to complete a 21-day cycle.
  Interventions: Drug: ABT-263
- Navitoclax 21/21 Day Cycle: 125 mg (Experimental): Navitoclax 125 mg administered for 21 consecutive days to complete a 21-day cycle.
  Interventions: Drug: ABT-263
- Navitoclax 21/21 Day Cycle: 200 mg (Experimental): Navitoclax 200 mg administered for 21 consecutive days to complete a 21-day cycle.
  Interventions: Drug: ABT-263
- Navitoclax 21/21 Day Cycle: 250 mg (Experimental): Navitoclax 250 mg administered for 21 consecutive days to complete a 21-day cycle.
  Interventions: Drug: ABT-263
- Navitoclax 21/21 Day Cycle: 300 mg (Experimental): Navitoclax 300 mg administered for 21 consecutive days to complete a 21-day cycle.
  Interventions: Drug: ABT-263
- Phase 2: Navitoclax 100 mg (Experimental): Navitoclax 100 mg in participants with CLL who had relapsed following any (but no more than 5) prior myelosuppressive/chemotherapy treatment regimen(s).
  Interventions: Drug: ABT-263
- Phase 2: Navitoclax 250 mg (Experimental): Navitoclax 250 mg in participants with CLL who had relapsed following any (but no more than 5) prior myelosuppressive/chemotherapy treatment regimen(s).
  Interventions: Drug: ABT-263

INTERVENTIONS:
Drug: ABT-263 — Tablet; Oral
  Other Names: Navitoclax

SUMMARY:
The Phase 1 portion of the study will evaluate the pharmacokinetic profile and safety of ABT-263 under two different dosing schedules with the objective of defining the dose limiting toxicity and maximum tolerated dose. The Phase 2a portion of the study will evaluate ABT-263 at the defined recommended Phase 2 dose to obtain additional safety information and a preliminary assessment of efficacy. The Extension Study portion will allow active subjects to continue to receive ABT-263 for up to 11 years after the last subject transitions with less frequent study evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory CLL and require treatment in opinion of investigator.
* Eastern Cooperative Oncology Group (ECOG) <= 1.
* Adequate bone marrow independent of growth factor support, renal and hepatic function per defined laboratory criteria.

Exclusion Criteria:

* History or is clinically suspicious for cancer-related Central Nervous System disease.
* Receipt of allogenic or autologous stem cell transplant.
* Recent history (within 1 year of first dose) of underlying, predisposing condition of bleeding or currently exhibits signs of bleeding.
* Active peptic ulcer disease or other potentially hemorrhagic esophagitis/gastritis.
* Active immune thrombocytopenic purpura or history of being refractory to platelet transfusions (within 1 year of first dose).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07-25 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (6):
  - Moores Cancer Center at UC San Diego /ID# 5566, La Jolla, California
  - Dana-Farber Cancer Institute /ID# 5547, Boston, Massachusetts
  - University of Nebraska Medical Center /ID# 12261, Omaha, Nebraska
  - North Shore University Hospital /ID# 12267, New Hyde Park, New York
  - University of Texas MD Anderson Cancer Center /ID# 5575, Houston, Texas
  - Northwest Medical Specialties - Tacoma /ID# 26428, Tacoma, Washington
- Australia (2):
  - Peter MacCallum Cancer Ctr /ID# 6583, Melbourne, Victoria
  - The Royal Melbourne Hospital /ID# 5576, Parkville, Victoria
- Universitaetsklinikum Koeln /ID# 5924, Cologne, North Rhine-Westphalia, Germany
- Leicester Royal Infirmary /ID# 15081, Leicester, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Result] Roberts AW, Seymour JF, Brown JR, Wierda WG, Kipps TJ, Khaw SL, Carney DA, He SZ, Huang DC, Xiong H, Cui Y, Busman TA, McKeegan EM, Krivoshik AP, Enschede SH, Humerickhouse R. Substantial susceptibility of chronic lymphocytic leukemia to BCL2 inhibition: results of a phase I study of navitoclax in patients with relapsed or refractory disease. J Clin Oncol. 2012 Feb 10;30(5):488-96. doi: 10.1200/JCO.2011.34.7898. Epub 2011 Dec 19. PMID 22184378
- See also: Related Info — https://www.abbvieclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 2: Navitoclax 100 mg: Navitoclax 100 mg in participants with chronic lymphocytic leukemia (CLL) who had relapsed following any (but no more than 5) prior myelosuppressive/chemotherapy treatment regimen(s).
Period: Overall Study
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg | Phase 2: Navitoclax 100 mg | Phase 2: Navitoclax 250 mg
Started | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4 | 4 | 27
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4 | 4 | 27
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 6
Not completed — Other, Not Specified | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Not completed — Adverse Event | 1 | 2 | 0 | 1 | 1 | 1 | 2 | 1 | 1 | 6
Not completed — Progressive disease clinical | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7
Not completed — Progressive disease clinical National Cancer Institute | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease other | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 0 | 0
Not completed — No reason given | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg | Phase 2: Navitoclax 100 mg | Phase 2: Navitoclax 250 mg | Total
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4 | 4 | 27 | 60
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 1 | 0 | 1 | 1 | 1 | 3 | 0 | 1 | 1 | 10 | 19
  >= 65 years | 2 | 6 | 2 | 2 | 2 | 1 | 3 | 3 | 3 | 17 | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 0 | 1 | 2 | 1 | 0 | 3 | 0 | 8 | 18
  Male | 1 | 5 | 3 | 2 | 1 | 3 | 3 | 1 | 4 | 19 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 6 | 2 | 3 | 2 | 3 | 2 | 3 | 4 | 24 | 52
  Black | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  American Indian/Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Mixed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Other, Not Specified | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 5
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  No Ethnicity | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4 | 4 | 27 | 60

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Discontinuations Due to Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An SAE is one that: results in death, hospitalization, prolongation of hospitalization, or persistent or significant disability/incapacity; is life-threatening, a congenital anomaly, or other important medical event. Events were graded as 1=mild, 2=moderate, 3=severe, 4=life-threatening, or 5=death. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A treatment-emergent adverse event is defined as any adverse event with onset or worsening reported by a subject from the time that the first dose of study drug is administered until 30 days have elapsed following discontinuation of study drug administration. Deaths category included non treatment emergent deaths.
Time Frame: From first dose of study drug to 30 days post-last dose. Participants enrolled in the 14/21-day cycle received a mean of 21.7 treatment cycles; participants enrolled in the 21/21-day cycle received a mean of 19.4 treatment cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4
Participants
  Any AE | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4
  Any AE at least possibly related to navitoclax | 3 | 4 | 3 | 3 | 3 | 4 | 3 | 4
  Any AE with NCI CTCAE Grade ≥ 3 | 2 | 4 | 3 | 2 | 2 | 4 | 3 | 4
  Any AE with NCI CTCAE Grade 3 or 4 | 2 | 4 | 3 | 2 | 2 | 4 | 3 | 4
  Any SAE | 2 | 4 | 2 | 2 | 2 | 4 | 2 | 3
  Any AE leading to navitoclax discontinuation | 1 | 2 | 0 | 1 | 2 | 1 | 2 | 1
  Any AE leading to navitoclax dose reduction | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 0
  Any AE leading to navitoclax interruption | 0 | 4 | 3 | 2 | 1 | 4 | 3 | 4
  Any AE leading to dose delay | 2 | 3 | 1 | 2 | 0 | 0 | 0 | 2
  Any dose limiting toxicity (DLT) | 0 | 2 | 0 | 2 | 0 | 2 | 2 | 2
  Any fatal AE | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Deaths | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0

2. Primary Outcome: Phase 1: Number of Participants With DLTs in the Dose Escalation Phase
Description: DLTs were graded according to NCI CTCAE version 3.0 (grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=life threatening; grade 5=death). Any of the following events, considered possibly or probably related to the administration of navitoclax, were considered a DLT: Grade 4 thrombocytopenia (< 25,000/mm^3); platelet counts < 25,000/mm^3, Grade 2 or higher bleeding associated with thrombocytopenia; all other Grade 3, 4 or 5 adverse events were considered a DLT. Exceptions included: Grade 3, 4 febrile neutropenia less than 7 days; Grade 3, 4 leukopenia; Grade 3, 4 lymphopenia; Grade 3 nausea, vomiting and/or diarrhea unless unresponsive to treatment; Grade 2 toxicity that requires dose modification or delay of > 1 week.
Time Frame: Cycle 1 (Up to 21 days) plus 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4
Participants | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1

3. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) in the Dose Escalation Phase
Description: The MTD was defined as the dose at which 30% of participants experienced a DLT during the first cycle. DLTs were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0 (grade 1=mild; grade 2=moderate; grade 3=severe; grade 4=life threatening; grade 5=death). Any of the following events, considered possibly or probably related to the administration of navitoclax, were considered a DLT: Grade 4 thrombocytopenia (< 25,000/mm^3); platelet counts < 25,000/mm^3, Grade 2 or higher bleeding associated with thrombocytopenia; all other Grade 3, 4 or 5 adverse events were considered a DLT. Exceptions included: Grade 3, 4 febrile neutropenia less than 7 days; Grade 3, 4 leukopenia; Grade 3, 4 lymphopenia; Grade 3 nausea, vomiting and/or diarrhea unless unresponsive to treatment; Grade 2 toxicity that requires dose modification or delay of > 1 week.
Time Frame: Cycle 1 (Up to 21 days) plus 7 days
Measure: Number; unit: mg
Groups:
- Participants Receiving 14/21-Day Dosing Schedule in Phase 1: Navitoclax 10, 110, 200, or 250 mg administered for 14 consecutive days followed by 7 days off drug to complete a 21-day cycle.
- Participants Receiving 21/21-Day Dosing Schedule in Phase 1: Navitoclax 125, 200, 250, or 300 mg administered for 21 consecutive days to complete a 21-day cycle.
Arm/Group | Participants Receiving 14/21-Day Dosing Schedule in Phase 1 | Participants Receiving 21/21-Day Dosing Schedule in Phase 1
Number analyzed (Participants) | 15 | 14
mg | 200 | 250

4. Primary Outcome: Phase 1: Recommended Phase 2 Dose (RPTD) Determined in the Dose Escalation Phase
Description: The RPTD was determined based on observed DLTs and/or determination of the MTD in phase 1. (See Outcome Measures 2 and 3 above for definition of DLT and MTD.)
Time Frame: Cycle 1 (Up to 21 days) plus 7 days
Measure: Number; unit: mg
Arm/Group | Participants Receiving 14/21-Day Dosing Schedule in Phase 1 | Participants Receiving 21/21-Day Dosing Schedule in Phase 1
Number analyzed (Participants) | 15 | 14
mg | 250 | 250

5. Primary Outcome: Phase 1: Time to Maximum Observed Plasma Concentration (Tmax) of Navitoclax
Time Frame: Cycle 1 Days 1 and 14: pre-dose, 2, 4, 6, 8 hours post-dose
Population: Participants with an assessment at given time point. One participant in the Navitoclax 14/21 Day Cycle: 250 mg arm dose-reduced to 200 mg on Days 4 to14, and therefore was analyzed in the Navitoclax 14/21 Day Cycle: 200 mg arm for Cycle 1 Day 14.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 3 | 4 | 3 | 4
hours
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4
  Cycle 1 Day 1 | 6.0 (2.0) | 5.9 (1.6) | 6.7 (1.2) | 7.3 (1.2) | 7.3 (1.2) | 6.5 (1.0) | 6.7 (2.3) | 7.5 (1.0)
  Cycle 1 Day 14: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 3 | 3 | 3
  Cycle 1 Day 14 | 4.3 (1.5) | 3.5 (2.8) | 6.8 (1.5) | 5.7 (0.4) | 5.8 (1.8) | 6.7 (1.2) | 6.9 (1.8) | 7.3 (1.2)

6. Primary Outcome: Phase 1: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Cycle 1 Days 1 and 14: pre-dose, 2, 4, 6, 8 hours post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 3 | 4 | 3 | 4
μg/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4
  Cycle 1 Day 1 | 0.25 (0.14) | 1.19 (0.37) | 2.60 (1.54) | 5.19 (2.70) | 2.24 (0.98) | 2.73 (0.82) | 2.59 (1.60) | 3.30 (1.20)
  Cycle 1 Day 14: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 3 | 3 | 3
  Cycle 1 Day 14 | 0.42 (0.17) | 1.87 (0.71) | 4.44 (3.59) | 3.21 (0.12) | 2.68 (1.11) | 3.46 (1.57) | 3.74 (1.19) | 3.11 (2.26)

7. Primary Outcome: Phase 1: Area Under the Plasma Concentration-Time Curve From Time 0 to Hour 8 (AUC8)
Time Frame: Cycle 1 Days 1 and 14: pre-dose, 2, 4, 6, 8 hours post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: μg•hr/mL
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 3 | 4 | 3 | 4
μg•hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 4 | 3 | 3 | 3 | 4 | 3 | 4
  Cycle 1 Day 1 | 1.0 (0.65) | 5.7 (2.7) | 10.6 (4.0) | 19.8 (14.0) | 12.0 (4.2) | 12.3 (3.0) | 12.0 (9.2) | 14.3 (5.7)
  Cycle 1 Day 14: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 3 | 3 | 3
  Cycle 1 Day 14 | 2.2 (0.95) | 11.1 (2.7) | 24.2 (18.1) | 17.8 (2.3) | 15.7 (6.8) | 18.4 (8.7) | 24.4 (5.7) | 21.6 (15.6)

8. Primary Outcome: Phase 1: Area Under the Plasma Concentration-Time Curve From Time 0 to Hour 24 (AUC24)
Description: The AUC24 was derived and reported from Cycle 1 Day 1 values and Cycle 1 Day 14 values; the pre-dose value taken on Day 14 was utilized as 24-hour timepoint on Day 14 to generate AUC24 for Day 14.
Time Frame: Cycle 1 Day 1: pre-dose, 2, 4, 6, 8, and 24 hours post-dose; Cycle 1 Days 14: pre-dose, 2, 4, 6, 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: μg•hr/mL
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 3 | 4 | 3 | 4
μg•hr/mL
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4
  Cycle 1 Day 1 | 2.7 (1.0) | 15.0 (3.2) | 34.0 (13.8) | 67.8 (27.7) | 37.5 (16.0) | 44.0 (18.7) | 49.5 (12.3) | 52.9 (20.1)
  Cycle 1 Day 14: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 3 | 3 | 3
  Cycle 1 Day 14 | 5.5 (2.7) | 30.9 (7.7) | 68.7 (42.9) | 50.6 (0.36) | 43.5 (16.6) | 56.2 (28.6) | 72.7 (14.4) | 64.8 (49.4)

9. Primary Outcome: Phase 1: Cmax/Dose
Time Frame: Cycle 1 Days 1 and 14: pre-dose, 2, 4, 6, 8 hours post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL/mg
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 3 | 4 | 3 | 4
ng/mL/mg
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4
  Cycle 1 Day 1 | 24.5 (13.9) | 10.7 (3.4) | 13.0 (7.7) | 20.8 (10.8) | 17.9 (7.9) | 13.7 (4.1) | 10.4 (6.4) | 11.0 (4.0)
  Cycle 1 Day 14: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 3 | 3 | 3
  Cycle 1 Day 14 | 42.3 (16.6) | 17.0 (6.4) | 22.2 (17.9) | 12.8 (0.48) | 21.4 (8.9) | 17.3 (7.9) | 15.0 (4.8) | 10.4 (7.5)

10. Primary Outcome: Phase 1: AUC8/Dose
Time Frame: Cycle 1 Days 1 and 14: pre-dose, 2, 4, 6, 8 hours post-dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng•hr/mL/mg
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 3 | 4 | 3 | 4
ng•hr/mL/mg
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4
  Cycle 1 Day 1 | 99.9 (65.0) | 52.0 (24.7) | 53.1 (20.1) | 79.2 (56.1) | 95.8 (33.5) | 61.3 (14.9) | 47.9 (36.8) | 47.6 (18.8)
  Cycle 1 Day 14: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 3 | 3 | 3
  Cycle 1 Day 14 | 215.0 (95.1) | 101.0 (24.7) | 121.0 (90.4) | 71.3 (9.1) | 125.0 (54.1) | 92.1 (43.3) | 97.7 (22.6) | 72.0 (51.9)

11. Primary Outcome: Phase 1: AUC24/Dose
Description: as for outcome 8
Time Frame: Cycle 1 Day 1: pre-dose, 2, 4, 6, 8, and 24 hours post-dose; Cycle 1 Days 14: pre-dose, 2, 4, 6, 8
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng•hr/mL/mg
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg
Number analyzed (Participants) | 3 | 6 | 4 | 3 | 3 | 4 | 3 | 4
ng•hr/mL/mg
  Cycle 1 Day 1: number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 4 | 3 | 4
  Cycle 1 Day 1 | 268 (100.0) | 136 (28.8) | 170 (69.2) | 271 (111.0) | 300 (128.0) | 220 (93.6) | 198 (49.3) | 176 (67.0)
  Cycle 1 Day 14: number analyzed (Participants) | 3 | 3 | 4 | 2 | 3 | 3 | 3 | 3
  Cycle 1 Day 14 | 546 (267.0) | 281 (69.9) | 344 (215.0) | 202 (1.5) | 348 (133.0) | 281 (143.0) | 291 (57.5) | 216.0 (165.0)

12. Primary Outcome: Phase 1: Terminal Phase Elimination Rate Constant (β) for Navitoclax
Time Frame: Cycle 1 Day 1: pre-dose, 2, 4, 6, 8 hours post-dose
Population: Participants with an assessment.
Measure: Mean (Standard Deviation); unit: 1/H
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg
Number analyzed (Participants) | 2 | 3 | 2 | 1 | 0 | 3 | 0 | 1
1/H | 0.072 (0.029) | 0.077 (0.006) | 0.067 (0.030) | 0.059 (NA) — not applicable (1 participant analyzed) |  | 0.066 (0.025) |  | 0.039 (NA) — not applicable (1 participant analyzed)

13. Primary Outcome: Phase 1: Terminal Phase Elimination Half-life (t1/2) of Navitoclax
Description: For t1/2, the harmonic mean and psuedo-standard deviation are used.
Time Frame: Cycle 1 Day 1: pre-dose, 2, 4, 6, 8 hours post-dose
Population: Participants with an assessment.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg
Number analyzed (Participants) | 2 | 3 | 2 | 1 | 0 | 3 | 0 | 1
hours | 9.62 (4.18) | 8.99 (0.66) | 10.41 (5.21) | 11.72 (NA) — Not applicable (1 participant analyzed) |  | 10.51 (4.01) |  | 17.88 (NA) — Not applicable (1 participant analyzed)

14. Primary Outcome: Phase 2: Number of Participants With TEAEs, SAEs, and Discontinuations Due to AEs
Description: as for outcome 1
Time Frame: From first dose of study drug to 30 days post-last dose. Participants enrolled in Phase 2 received a mean of 15.6 treatment cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Navitoclax 100 mg | Phase 2: Navitoclax 250 mg
Number analyzed (Participants) | 4 | 27
Participants
  Any AE | 4 | 27
  Any AE at least possibly related to navitoclax | 4 | 26
  Any AE with NCI CTCAE Grade ≥ 3 | 3 | 23
  Any AE with NCI CTCAE Grade 3 or 4 | 3 | 23
  Any SAE | 1 | 12
  Any AE leading to navitoclax discontinuation | 1 | 9
  Any AE leading to navitoclax dose reduction | 1 | 10
  Any AE leading to navitoclax interruption | 2 | 16
  Any AE leading to navitoclax dose delay | 2 | 5
  Any fatal AE | 0 | 1
  Deaths | 1 | 8

15. Primary Outcome: Phase 2: Dose-Normalized Plasma Concentrations After Navitoclax Once Daily Dosing
Time Frame: Cycle 1 Day 1: 4-8 h postdose; Cycle 1 Day 15: predose; Cycle 3 Day 1: predose, 4-8 h postdose; Cycle 5 Day 1: predose, 4-8 h postdose; Cycle 7 Day 1: predose, 4-8 h postdose; Cycle 9 Day 1: predose, 4-8 h postdose
Population: Participants with an assessment at given time point. It was pre-specified in the statistical analysis plans to analyze the dose-normalized assessments in phase 2 navitoclax arms combined.
Measure: Mean (Standard Deviation); unit: (ng/mL)/mg
Groups:
- Participants Receiving Navitoclax QD Dosing in Phase 2: Navitoclax 100 mg or 250 mg in participants with CLL who had relapsed following any (but no more than 5) prior myelosuppressive/chemotherapy treatment regimen(s).
Arm/Group | Participants Receiving Navitoclax QD Dosing in Phase 2
Number analyzed (Participants) | 31
(ng/mL)/mg
  Cycle 1 Day 1: 4-8 h postdose: number analyzed (Participants) | 25
  Cycle 1 Day 1: 4-8 h postdose | 9.49 (4.80)
  Cycle 1 Day 15: predose: number analyzed (Participants) | 22
  Cycle 1 Day 15: predose | 9.64 (5.85)
  Cycle 3 Day 1: predose: number analyzed (Participants) | 20
  Cycle 3 Day 1: predose | 9.84 (3.55)
  Cycle 3 Day 1: 4-8 h postdose: number analyzed (Participants) | 17
  Cycle 3 Day 1: 4-8 h postdose | 15.2 (8.04)
  Cycle 5 Day 1: predose: number analyzed (Participants) | 21
  Cycle 5 Day 1: predose | 9.84 (4.38)
  Cycle 5 Day 1: 4-8 h postdose: number analyzed (Participants) | 19
  Cycle 5 Day 1: 4-8 h postdose | 15.7 (8.28)
  Cycle 7 Day 1: predose: number analyzed (Participants) | 9
  Cycle 7 Day 1: predose | 10.4 (5.26)
  Cycle 7 Day 1: 4-8 h postdose: number analyzed (Participants) | 9
  Cycle 7 Day 1: 4-8 h postdose | 15.9 (9.14)
  Cycle 9 Day 1: predose: number analyzed (Participants) | 5
  Cycle 9 Day 1: predose | 11.4 (9.68)
  Cycle 9 Day 1: 4-8 h postdose: number analyzed (Participants) | 4
  Cycle 9 Day 1: 4-8 h postdose | 13.5 (6.41)

ADVERSE EVENTS:
Time Frame: Adverse events: From first dose of study drug to 30 days post-last dose. Participants enrolled in the 14/21-day cycle received a mean of 21.7 treatment cycles; participants enrolled in the 21/21-day cycle received a mean of 19.4 treatment cycles. Participants enrolled in Phase 2 received a mean of 15.6 treatment cycles.
Description: Time frame for All Cause Mortality: From informed consent to the end of study. Median time on study: 135, 89.5, 608, 441, 299, 307, 561, 152.5, 486.5, 803 days for Ph 1 14/21 Day Cycle 10 mg, 110 mg, 200 mg, 250 mg, Ph 1 21/21 Day Cycle 125 mg, 200 mg, 250 mg, 300mg and Ph 2 100 mg , 250 mg arms, respectively.
Groups:
- Navitoclax 14/21 Day Cycle: 10 mg: Navitoclax 10 mg administered for 14 consecutive days followed by 7 days off drug to complete a 21- day cycle.
- Navitoclax 14/21 Day Cycle: 110 mg: Navitoclax 110 mg administered for 14 consecutive days followed by 7 days off drug to complete a 21- day cycle.
- Navitoclax 14/21 Day Cycle: 200 mg: Navitoclax 200 mg administered for 14 consecutive days followed by 7 days off drug to complete a 21- day cycle.
- Navitoclax 14/21 Day Cycle: 250 mg: Navitoclax 250 mg administered for 14 consecutive days followed by 7 days off drug to complete a 21- day cycle.
- Phase 2: Navitoclax 100 mg: Navitoclax 100 mg in subjects with CLL who had relapsed following any (but no more than 5) prior myelosuppressive/chemotherapy treatment regimen(s).
- Phase 2: Navitoclax 250 mg: Navitoclax 250 mg in subjects with CLL who had relapsed following any (but no more than 5) prior myelosuppressive/chemotherapy treatment regimen(s).
Arm/Group | Navitoclax 14/21 Day Cycle: 10 mg | Navitoclax 14/21 Day Cycle: 110 mg | Navitoclax 14/21 Day Cycle: 200 mg | Navitoclax 14/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 125 mg | Navitoclax 21/21 Day Cycle: 200 mg | Navitoclax 21/21 Day Cycle: 250 mg | Navitoclax 21/21 Day Cycle: 300 mg | Phase 2: Navitoclax 100 mg | Phase 2: Navitoclax 250 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/6 | 0/3 | 0/3 | 1/3 | 0/4 | 0/3 | 0/4 | 1/4 | 8/27
Serious Adverse Events (participants affected / at risk) | 2/3 | 4/6 | 2/3 | 2/3 | 2/3 | 4/4 | 2/3 | 3/4 | 1/4 | 12/27
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 3/3 | 3/3 | 3/3 | 4/4 | 3/3 | 4/4 | 4/4 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navitoclax 14/21 Day Cycle: 10 mg (N=3) | Navitoclax 14/21 Day Cycle: 110 mg (N=6) | Navitoclax 14/21 Day Cycle: 200 mg (N=3) | Navitoclax 14/21 Day Cycle: 250 mg (N=3) | Navitoclax 21/21 Day Cycle: 125 mg (N=3) | Navitoclax 21/21 Day Cycle: 200 mg (N=4) | Navitoclax 21/21 Day Cycle: 250 mg (N=3) | Navitoclax 21/21 Day Cycle: 300 mg (N=4) | Phase 2: Navitoclax 100 mg (N=4) | Phase 2: Navitoclax 250 mg (N=27)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AMOEBIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPERGILLUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
GASTROENTERITIS SALMONELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROGRESSIVE MULTIFOCAL LEUKOENCEPHALOPATHY (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COLORECTAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT MELANOMA OF EYELID (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUPERFICIAL SPREADING MELANOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TRANSIENT ISCHEMIC ATTACK (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navitoclax 14/21 Day Cycle: 10 mg (N=3) | Navitoclax 14/21 Day Cycle: 110 mg (N=6) | Navitoclax 14/21 Day Cycle: 200 mg (N=3) | Navitoclax 14/21 Day Cycle: 250 mg (N=3) | Navitoclax 21/21 Day Cycle: 125 mg (N=3) | Navitoclax 21/21 Day Cycle: 200 mg (N=4) | Navitoclax 21/21 Day Cycle: 250 mg (N=3) | Navitoclax 21/21 Day Cycle: 300 mg (N=4) | Phase 2: Navitoclax 100 mg (N=4) | Phase 2: Navitoclax 250 mg (N=27)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (7)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 2 (5) | 0 (0) | 7 (20)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (10) | 2 (10) | 0 (0) | 1 (5) | 0 (0) | 1 (3) | 1 (2) | 13 (39)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PHIMOSIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR CONGESTION (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EAR DISCOMFORT (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
AUTOIMMUNE HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DACRYOSTENOSIS ACQUIRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECTROPION (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EYE HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SWELLING OF EYELID (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (6)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 2 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (2) | 4 (9) | 3 (15) | 3 (4) | 2 (8) | 3 (6) | 3 (10) | 3 (9) | 4 (5) | 20 (30)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 3 (4) | 2 (8) | 2 (2) | 3 (6) | 2 (6) | 2 (2) | 2 (2) | 2 (2) | 13 (17)
NONINFECTIVE GINGIVITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
RECTAL FISSURE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RECTAL POLYP (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
TONGUE ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 2 (9) | 2 (3) | 1 (2) | 1 (1) | 1 (1) | 5 (5)
ADVERSE DRUG REACTION (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST DISCOMFORT (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 0 (0) | 3 (7) | 2 (4) | 2 (2) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 1 (2) | 10 (14)
FEELING HOT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OEDEMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 7 (7)
PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (5)
SECRETION DISCHARGE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VESSEL PUNCTURE SITE PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4)
ALLERGY TO ARTHROPOD BITE (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ACUTE SINUSITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ESCHERICHIA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
EYE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAEMOPHILUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HERPES SIMPLEX (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LICE INFESTATION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOCALISED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 2 (5) | 1 (4) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 5 (7)
ORAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOOTH ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 2 (5) | 1 (6) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 8 (11)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 1 (5) | 0 (0) | 5 (10)
VASCULAR DEVICE INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUNBURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (9) | 0 (0) | 1 (2) | 3 (6)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
BLOOD MAGNESIUM DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5)
HEART RATE IRREGULAR (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 3 (3)
WEIGHT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 1 (1) | 8 (10)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (6)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
OSTEITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
COLORECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APHASIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (4)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 3 (4)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SENSORY DISTURBANCE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TASTE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
INSOMNIA (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL CYST (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RENAL PAIN (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PENILE CURVATURE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROSTATITIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (4) | 1 (1) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 6 (7)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 1 (1) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 3 (5)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SPUTUM DISCOLOURED (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
BLOOD BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DERMATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3)
RASH VESICULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN DISCOLOURATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
VASCULITIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/91/NCT00481091/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-27): https://cdn.clinicaltrials.gov/large-docs/91/NCT00481091/SAP_001.pdf